CLINICAL TRIAL: NCT00722865
Title: Avastin (Bevacizumab) in Combination With ABVD for the Treatment of Newly Diagnosed Advanced Stage Classical Hodgkin Lymphoma
Brief Title: Avastin (Bevacizumab) Plus Adriamycin, Bleomycin, Vinblastine and Dacarbazine (ABVD) for Advanced Stage Hodgkin Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Jeremy Abramson, MD, Director, Lymphoma Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-388
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Results first posted 2017-04-28 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-09

CONDITIONS: Hodgkin Lymphoma
Keywords: Avastin; bevacizumab; ABVD; angiogenesis; antiangiogenic; Hodgkin
MeSH Terms: conditions — Hodgkin Disease | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avastin (Bevacizumab) (Other): single-arm, open-label
  Interventions: Drug: Avastin

INTERVENTIONS:
Drug: Avastin — Given intravenously along with standard chemotherapy (Adriamycin, Bleomycin, Vinblastine and Dacarbazine) on days 1 and 15 of a 28-day cycle for a total of 6 planned cycles.
  Other Names: Bevacizumab

SUMMARY:
The purpose of this research study is to determine the effectiveness and safety of Avastin when combined with standard chemotherapy for Hodgkin lymphoma. Avastin works differently than standard chemotherapy drugs. It is a type of protein called an antibody which binds to a substance called VEGF(Vascular Endothelial Growth Factor). VEGF stimulates the growth of the blood vessels that feed tumors and encourages tumor cell growth. VEGF is produced in excess by Hodgkin lymphoma cells, and is associated with a poorer outcome in patients with Hodgkin lymphoma. When the activity of VEGF is interrupted in multiple other cancer types, the blood vessels around the tumor cells die resulting in less nutrient delivery and death to the tumor. Blocking of VEGF has also been shown to improve delivery of chemotherapy to cancer cells, making standard chemotherapy work better. This trial uses Avastin in combination with standard chemotherapy with the goal of improving the cure rate over chemotherapy alone.

DETAILED DESCRIPTION:
Participants will be given Avastin as well as ABVD (Adriamycin, Bleomycin, Vinblastine and Dacarbazine) intravenously on days 1 and 15 of a 28 day cycle. Participants will receive up to a total of 6 cycles of therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Biopsy proven classical Hodgkin lymphoma. Classical Hodgkin lymphoma includes the subtypes of nodular sclerosis, mixed cellularity, lymphocyte rich, lymphocyte depleted, and classical Hodgkin lymphoma unspecified
* Advanced stage (Stage III or IV) disease
* Measurable disease on cross sectional imaging
* ECOG Performance Status 0-2
* Adequate blood counts and organ function

Exclusion Criteria:

* Pregnant or lactating women
* Laboratory Parameters as outlined in the protocol
* LV ejection fraction lower than normal as assessed by echocardiogram or MUGA scan
* DLCO less than 60% as measured by pulmonary function tests
* Prior history of another malignancy (except for non-melanoma skin cancer or in situ cervical or breast cancer) unless disease free for over one year
* Current or recent (within 4 weeks of the first infusion of this study) participation in an experimental drug study
* Life expectancy of less than 12 weeks
* Inability to comply with study procedures
* Inability to give informed consent
* Inadequately controlled hypertension
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* NYHA Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Known CNS involvement of Hodgkin lymphoma
* Significant vascular disease
* Symptomatic peripheral vascular disease
* Evidence of bleeding diatheses or coagulopathy
* Use of daily anticoagulant medications including warfarin, heparins, or aspirin >325mg daily
* Major surgical procedure or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days of study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening
* Known hypersensitivity to any component of bevacizumab
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Abramson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Avastin (Bevacizumab)
Started | 25
Completed | 23
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Avastin (Bevacizumab)
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 29 [18 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 25
Stage of Cancer [Count of Participants; unit: Participants]
  Stage III | 10
  Stage IV | 15
Hemoglobin [Count of Participants; unit: Participants]
  <10.5 g/dL | 7
  >=10.5 g/dL | 18
Leukocytosis [Count of Participants; unit: Participants]
  >15,000/uL | 5
  <=15,000/uL | 20
Absolute lymphocyte count [Count of Participants; unit: Participants]
  <600/uL | 4
  >=600/uL | 21
Albumin [Count of Participants; unit: Participants]
  <4.0 g/dL | 17
  >=4.0 g/dL | 8
B symptoms [Count of Participants; unit: Participants] — B symptoms refer to systemic symptoms of fever, night sweats, and weight loss which can be associated with both Hodgkin's lymphoma and non-Hodgkin's lymphoma. The presence or absence of B symptoms has prognostic significance and is reflected in the staging of these lymphomas.
  Participants
    Yes | 15
    No | 10
International Prognostic Scoring System (IPSS) [Count of Participants; unit: Participants] — Risk score: 0-1= very low, 2 = low, 3 = intermediate, 4-5=high
  Participants
    0 | 1
    1 | 5
    2 | 5
    3 | 4
    4 | 7
    5 | 3

OUTCOME MEASURES:

1. Primary Outcome: Failure-free Survival
Description: Failure-free survival: the absence of relapse, non-relapse mortality or addition of another systemic therapy
Time Frame: 2 years and median follow-up of 18 months
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Avastin (Bevacizumab)
Number analyzed (Participants) | 25
percentage of participants
  at 2 years | 67 [50 to 84]
  at median follow-up of 18 months | 73 [57 to 88]

2. Secondary Outcome: Overall Response Rate Using the Modified Cheson Criteria
Description: Overall response = Complete response (CR) + Partial response (PR) CR = all previously enlarged fluorodeoxyglucose (FDG)-avid or positron emission tomography (PET)-positive lymph nodes regressed to normal size (<=1.5cm in greatest diameter) PR = >=50% decrease in SPD of up to six largest dominant masses, no increase in size of other nodes; FDG avid or PET positive before therapy, one or more nodes PET positive at previously involved site, or variably FDG avid or PET negative with regression at CT
Time Frame: 2 years
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Avastin (Bevacizumab)
Number analyzed (Participants) | 25
percentage of participants | 96 [82 to 99]

3. Secondary Outcome: Progression-free Survival
Description: Progression-free survival: a patient lives with the disease but it does not get worse.
Time Frame: 2 years and medium follow-up of 18 months
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Avastin (Bevacizumab)
Number analyzed (Participants) | 25
percentage of participants
  at 2 years | 67 [50 to 84]
  at median follow-up of 18 months | 73 [57 to 88]

4. Secondary Outcome: Overall Survival
Description: Overall survival: patients are still alive.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Avastin (Bevacizumab)
Number analyzed (Participants) | 25
Participants | 25

5. Secondary Outcome: Safety
Description: Toxicities are graded 1 (mild), 2 (moderate), 3 (severe), and 4 (life-threatening)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Avastin (Bevacizumab)
Number analyzed (Participants) | 25
Participants
  Anemia: Grade 1-2 | 19
  Anemia: Grade 3-4 | 3
  Anemia: Did not have any | 3
  Neutropenia: Grade 1-2 | 1
  Neutropenia: Grade 3-4 | 22
  Neutropenia: Did not have any | 2
  Thrombocytopenia: Grade 1-2 | 3
  Thrombocytopenia: Grade 3-4 | 0
  Thrombocytopenia: Did not have any | 22
  Febrile neutropenia: Grade 1-2 | 0
  Febrile neutropenia: Grade 3-4 | 4
  Febrile neutropenia: Did not have any | 21
  Hypertension: Grade 1-2 | 2
  Hypertension: Grade 3-4 | 1
  Hypertension: Did not have any | 22
  Proteinuria: Grade 1-2 | 0
  Proteinuria: Grade 3-4 | 0
  Proteinuria: Did not have any | 25
  Pericardial effusion: Grade 1-2 | 1
  Pericardial effusion: Grade 3-4 | 1
  Pericardial effusion: Did not have any | 23
  Pleural effusion: Grade 1-2 | 1
  Pleural effusion: Grade 3-4 | 0
  Pleural effusion: Did not have any | 24
  Skin breakdown: Grade 1-2 | 0
  Skin breakdown: Grade 3-4 | 1
  Skin breakdown: Did not have any | 24
  Mucositis: Grade 1-2 | 4
  Mucositis: Grade 3-4 | 0
  Mucositis: Did not have any | 21
  Sensory neuropathy: Grade 1-2 | 8
  Sensory neuropathy: Grade 3-4 | 1
  Sensory neuropathy: Did not have any | 16
  Thrombosis/embolism: Grade 1-2 | 0
  Thrombosis/embolism: Grade 3-4 | 2
  Thrombosis/embolism: Did not have any | 23
  Renal failure: Grade 1-2 | 0
  Renal failure: Grade 3-4 | 1
  Renal failure: Did not have any | 24
  Fatigue: Grade 1-2 | 21
  Fatigue: Grade 3-4 | 1
  Fatigue: Did not have any | 3

ADVERSE EVENTS:
Arm/Group | Avastin (Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 4/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin (Bevacizumab) (N=25)
Sensory Neuropathy (Nervous system disorders) | 1 (1) — grade 4, expected and definitely related
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) — grade 4, possibly related, expected
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — grade 4, possibly related, expected
Pericardial Effusion (Cardiac disorders) | 1 (1) — grade 3, possibly related, expected
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin (Bevacizumab) (N=25)
Ascites (Gastrointestinal disorders) | 25 (165)
Platelets (Blood and lymphatic system disorders) | 25 (165)
Chills (General disorders) | 25 (165)
Febrile neutropenia (Blood and lymphatic system disorders) | 25 (165)
Vomiting (Gastrointestinal disorders) | 25 (165)
Leukocytosis (Blood and lymphatic system disorders) | 25 (165)
Head/headache (General disorders) | 25 (165)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 25 (165)
Jejunal fistula (Gastrointestinal disorders) | 25 (165)
Pain of skin (Skin and subcutaneous tissue disorders) | 25 (165)
Anal hemorrhage (Gastrointestinal disorders) | 14 (25)
Movements involuntary (Nervous system disorders) | 9 (23)
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 7 (11)
Abdomen- pain (General disorders) | 5 (12)
Back- pain (General disorders) | 5 (12)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (14)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Anorectal infection (Infections and infestations) | 4 (6)
Edema face (General disorders) | 4 (5)
Gastritis (Gastrointestinal disorders) | 4 (5)
Extremity-limb- pain (General disorders) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 3 (8)
Nose- hemorrhage (Blood and lymphatic system disorders) | 3 (7)
Conduction disorder (Cardiac disorders) | 3 (5)
Hypertension (Cardiac disorders) | 3 (5)
Death neonatal (General disorders) | 3 (5)
Ileal obstruction (Gastrointestinal disorders) | 3 (5)
Edema cerebral (Nervous system disorders) | 3 (5)
Periorbital edema (Skin and subcutaneous tissue disorders) | 3 (4)
Neck- pain (General disorders) | 3 (3)
Pericardial effusion (non-malignant) (Cardiac disorders) | 2 (8)
Alkalosis (Metabolism and nutrition disorders) | 2 (7)
Fatigue (General disorders) | 2 (3)
Infection Gr0-2 neut, upper airway (Infections and infestations) | 2 (3)
Joint, pain (General disorders) | 2 (3)
Pain-other (General disorders) | 2 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Myocarditis (Cardiac disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Wound infection (Infections and infestations) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Chest wall, pain (General disorders) | 2 (2)
Throat/pharynx/larynx- pain (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No